CLINICAL TRIAL: NCT03995394
Title: Use of Text Messaging for Positive Reinforcement to Help Improve Quality of Life in Pediatric Obese Patients
Brief Title: Text Messaging Pediatric Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marsha Ma (Other)
Responsible Party: Sponsor-Investigator, Marsha Ma, Principal Investigator, Loyola University
Organization: Loyola University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 211950
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Reinforcement Group (Experimental): In the intervention group, participants will receive two text messages weekly. The first text message will ask if participants completed the recommended activity. If the participants respond yes, the participant will receive a positive reinforcement response. If the participants respond no, the participant will receive a text message stating, "Thank you for your response."
  Interventions: Other: Positive Reinforcement Text Message
- Control Group (No Intervention): For the control group, participants will receive two text messages weekly. The first text message will ask if the participants completed the recommended activity. When the participant responds, the participant will receive a second text message stating, "Thanks for your response."

INTERVENTIONS:
Other: Positive Reinforcement Text Message — A text message comprising the words, "Great job! We're so proud of you! Keep up the good work!"
  Arms: Positive Reinforcement Group

SUMMARY:
This study hopes to investigate the relationship between positive reinforcement for exercise activities in pediatric obese participants and quality of life. The investigators hypothesize that providing positive reinforcement through text messaging to children living with obesity will improve their overall quality of life. The investigators will recruit pediatric obese participants and administer a pre and post survey regarding quality of life. The family will be given recommendations on various ways to increase physical activity weekly. These participants will then receive positive reinforcement for completed exercises through text messages.

DETAILED DESCRIPTION:
This will be a prospective interventional cohort study following a group of participants with obesity. Informed consent will be obtained from the parents from a member of the research committee. Informed assent will also be obtained from the participant from a member of the research committee.

The investigators will review the schedule in the pediatrics department daily and approach all participants that meet our inclusion criteria. Per standard of care for participants with obesity, the participants have a scheduled follow up for a weight check at regular intervals that can include one month, 3 months or 6 months.

The 40 participants will be randomly assigned to either a control group or an intervention group.

Survey:

A 23 item PedsQL 4.0 pre-survey will be administered to pediatric participants to establish a baseline at their wellness visits. The parent of the participant will also be given a PedsQL survey to fill out. The participants' Body Mass Index (BMI) and blood pressure will be recorded. At the end of the 6-month period, the same PedsQL 4.0 will be administered again to both the participant and parent at the scheduled 6-month weight check that is standard of care.

The investigators will use a text message application created by the Loyola informatics team. This application will be able to text the participants using their cell phone number via an email service from the provider. For example, 123456789@cellservice provider.com. This allows the research team to send text messages to be sent through an application without using a personal phone number. In addition, it offers automatic responses that will save them when sending messages to the participant.

For six months, participants in the study will receive a text message twice per week via this application.

Text messaging:

There will be two groups within this study-a control group and an intervention group. For the control group, participants will receive two text messages weekly. The first text message will ask if the participants have completed the recommended activity. When a participant responds, the participant will receive a second text message stating, "Thanks for your response."

In the intervention group, the first text message will ask if the participant completed the recommended activity. If the participant responds yes, the participant will receive a positive reinforcement response comprising the words "Great job! We're so proud of you! Keep up the good work!". If the participant responds no, the participant will receive a text message stating, "Thank you for your response."

Study Activities:

The weekly activities the investigators will recommend for the participants include:

1. Walking for 30 minutes 3 times a week
2. Speed walk for 30 minutes 3 times a week
3. Walk up and down stairs for 30 minutes 3 times a week
4. Jogging for 30 minutes 3 times a week
5. Jumping jacks for 30 minute 3 times a week

Data:

All participant data will be stored in a protected Data-base, REDcap.

Statistical analysis:

In this study, participants who are age 18 and under with a BMI in at least the 95th percentile will be asked to complete assigned exercises. For six months, these participants will receive a text message twice per week asking whether the participant has completed the assigned exercises. For participants marking "Yes", exactly one half will be randomized to receive a positive reinforcement response comprising the words "Great job! We're so proud of you! Keep up the good work!". The other half will receive a control response comprising the words "Thanks for your response"; all participants marking "No" will receive this same response. The study will use a 1:1 allocation.

Six months following randomization, one goal of the proposed study is to test the null hypothesis that average total score on PedsQL 4.0 questionnaire between the two groups are equal. With a proposed sample size of 20 assigned to receive the positive reinforcement response and 20 assigned to receive the control response (N = 40), the study will have power of 80.0 percent to yield a statistically significant result. This computation assumes a mean difference between the two cohorts of 14.8 points (corresponding to means of 81.8 for the positive reinforcement cohort and 67.0 for the control response cohort) and a common within-group standard deviation of 16.3 points (Schwimmer, et al.). This computation also assumes the criterion for significance (alpha) is 0.05 and that the test will be 2-tailed, meaning an effect in either direction will be interpreted.

Recommended Protocol Text for the Analysis Plan:

Participants under age 18 with a BMI in at least the 95th percentile will be asked to complete assigned exercises and will receive text messages asking the participants if the participant has completed such exercises. At baseline and the end of the study, the participants will complete the 23-item PedsQL 4.0 assessment. For each participant, the baseline value will be subtracted from the 6-month value. An independent samples t-test will be used to compare this delta score between the cohort assigned to receive the positive reinforcement response and the cohort assigned to receive the control response. For this comparison, the normal distribution assumption of the delta score will be assessed using QQ plots and outliers will be assessed using box plots. The homogeneity of variances assumption will be assessed using Levene's test. If any parametric assumption is strongly violated, a non-parametric Wilcoxon rank-sum test may be used to compare ranked PedsQL 4.0 scores between the two cohorts. All analyses will be completed using SAS version 9.4 (Cary, NC) by a Biostatistician in the Clinical Research Office.

Safety Monitoring Plan:

There are no adverse events that could be associated with text messages the investigators will send to the participants. The investigators will send these text messages on Monday early evening between the 5pm to 6pm. The investigators chose this time because participants will not be in school and are unlikely to be driving or doing activities that the participants could be distracted from when receiving the text, which could cause harm.

If there is an adverse effect, the investigators will ask the participants to notify the principal investigator of the project. The investigators will review safety information once a month.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >95th percentile
* Has a cell phone

Exclusion Criteria:

* Developmental delay and inability to read
* Does not have a cell phone

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Pediatric Quality of Life Inventory 4.0 (PedsQL) Survey (child self-report 13-18) at 6 Months | 6-month
  This is a measurement of the participant's reported health-related quality of life while living with pediatric obesity. It is a multidimensional, 23-item survey measuring core elements of health, physical, emotional, social, and school functioning. The survey is a 5-point Likert scale from 0 (Never) to 4 (Almost always) and the scores are transformed on a scale from 0-100 as follows: 0=100, 1=75, 2=50, 3=25, 4=0. The mean score is the sum of the items over the number of items answered. The total score is the sum of all the items over the number of items answered on all the scales. Higher scores will indicate better health related quality of life. Lower scores will indicate worse health related quality of life.

SECONDARY OUTCOMES:
Mean Change from Baseline in Pediatric Quality of Life Inventory 4.0 (PedsQL) Survey (parent proxy report 13-18) at 6 Months | 6-month
  This is a measurement of the parent's perspective of the health-related quality of life of their child living with pediatric obesity. It is a multidimensional, 23-item survey measuring core elements of health, physical, emotional, social, and school functioning. The survey is a 5-point Likert scale from 0 (Never) to 4 (Almost always) and the scores are transformed on a scale from 0-100 as follows: 0=100, 1=75, 2=50, 3=25, 4=0. The mean score is the sum of the items over the number of items answered. The total score is the sum of all the items over the number of items answered on all the scales. Higher scores will indicate better health related quality of life. Lower scores will indicate worse health related quality of life.
Mean Change from Baseline in Body Mass Index (BMI) | 6-month
  This is a measurement of the participant's scheduled 6 month weight check that is the standard of care in pediatric obese patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Ma, M.D., Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwimmer JB, Burwinkle TM, Varni JW. Health-related quality of life of severely obese children and adolescents. JAMA. 2003 Apr 9;289(14):1813-9. doi: 10.1001/jama.289.14.1813. PMID 12684360

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03995394/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03995394/ICF_000.pdf